CLINICAL TRIAL: NCT00564070
Title: CBT for Adherence and Depression in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven A. Safren, Director, Behavioral Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH078571 (NIH); R01MH078571 (NIH)
Record Dates: First submitted 2007-11-23; First posted 2007-11-27 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus; Depression
Keywords: Depression; Diabetes; Adherence
MeSH Terms: conditions — Diabetes Mellitus; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced treatment as usual (Active Comparator): Enhanced treatment as usual plus single-session life-steps treatment
  Interventions: Behavioral: Enhanced treatment as usual plus adherence training
- CBT-AD (Experimental): Enhanced treatment as usual plus multiple-session CBT treatment (CBT-AD)
  Interventions: Behavioral: Enhanced treatment as usual plus CBT-AD

INTERVENTIONS:
Behavioral: Enhanced treatment as usual plus adherence training — The single-session life-steps treatment targets informational, problem solving, and cognitive-behavioral steps that are geared toward improving medication adherence and diabetes self-management.
  Arms: Enhanced treatment as usual
Behavioral: Enhanced treatment as usual plus CBT-AD — The multiple-session CBT treatment is given after completion of the life-steps session. The CBT sessions focus on treatment of depressive symptoms as well as adherence to diabetes self-care.
  Arms: CBT-AD

SUMMARY:
This study will evaluate the effectiveness of cognitive behavioral therapy (CBT) in treating people with depression and type 2 diabetes.

DETAILED DESCRIPTION:
Depression is a serious illness that affects a person's mood, thoughts, and physical being. Common symptoms of depression include persistent feelings of anxiety, guilt, or hopelessness; irregular sleep and appetite patterns; lethargy; disinterest in previously enjoyed activities; excessive irritability and restlessness; suicidal thoughts; and inability to concentrate. Depression is highly comorbid, often occurring in the presence of one or more other disorders. Up to 15% to 20% of the time, people with diabetes are also depressed. Diabetes is a disease that interferes with the body's proper production and use of the hormone insulin, which is needed to convert food into the energy required to perform daily life activities. Self-care is a crucial component of diabetes treatment. However, symptoms of depression can interfere with behaviors necessary to carry out this care. Cognitive behavioral therapy (CBT) has shown success in treating people with depression, but the effect of CBT on self-care behaviors and depression of those with diabetes is not well known. This study will evaluate the effectiveness of CBT for medical adherence and depression (CBT-AD) in people with a depressive mood disorder and type 2 diabetes.

Upon study entry, all participants will complete various assessments, including a psychiatric diagnostic interview, a series of paper questionnaires, neuropsychological testing, blood sample analysis, and blood sugar monitoring. Next, all participants will meet with a nutritionist and a nurse diabetes educator. The nutritionist will help set goals for eating, physical activity, weight, and blood glucose. The nurse diabetes educator will review diabetes medication history and blood glucose self-monitoring equipment.

Participants will then be randomly placed in one of two counseling groups. One group will meet for a single session that will be devoted to diabetes medical adherence. The other group will attend 10 to12 individual CBT sessions for diabetes medical adherence and depression management. The CBT sessions will last 45 to 50 minutes and will require practice of coping skills outside the sessions. Participants receiving CBT will also complete weekly assessments of depression, self-care, and diabetes medical adherence. All participants will be asked to monitor a prescribed medication with a pill cap for the course of the study. At Month 2, participants in both groups will also meet again with the nutritionist to review original goals and adjust them as necessary. Most of the previous study assessments will be repeated at Months 4, 8, and 12. The neuropsychological testing will be repeated only at Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes that is poorly controlled despite treatment with an oral hypoglycemic, insulin, or both
* Diagnosis of major depression or dysthymia, or current subclinical symptoms of depression in spite of prescription of an antidepressant
* If on an antidepressant, oral hypoglycemic medication, or insulin, must have been on a stable dose for the preceding two months

Exclusion Criteria:

* Active untreated major mental illness (e.g., untreated psychosis), bipolar disorder, eating disorder, mental retardation, or dementia
* Experiencing suicidal thoughts
* History of or currently receiving CBT for depression
* Uses an insulin pump

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Psaros, PhD, Study Director — Partners HealthCare; Steven Safren, PhD, Principal Investigator — University of Miami
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Safren SA, Gonzalez JS, Wexler DJ, Psaros C, Delahanty LM, Blashill AJ, Margolina AI, Cagliero E. A randomized controlled trial of cognitive behavioral therapy for adherence and depression (CBT-AD) in patients with uncontrolled type 2 diabetes. Diabetes Care. 2014;37(3):625-33. doi: 10.2337/dc13-0816. Epub 2013 Oct 29. PMID 24170758

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Started | 42 | 45
Completed | 30 | 38
Not Completed | 12 | 7
Not completed — Lost to Follow-up | 9 | 7
Not completed — Worsening depression, referred to care | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Treatment as Usual | CBT-AD | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.31 (7.41) | 55.44 (8.72) | 56.87 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 34 | 38 | 72
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 39 | 45 | 84
  Unknown or Not Reported | 0 | 0 | 0
Clinician-Rated Depression [Mean (Standard Deviation); unit: units on a scale] — Depression as assessed by the Montgomery Asberg Depression Rating Scale (MADRS). This scale has a range of 0-60 with higher scores indicating greater depression severity.
  units on a scale | 23.31 (7.20) | 25.60 (8.99) | 24.46 (8.10)
HbA1C [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — Hemoglobin A1C value at acute outcome. HbA1c is the number of hemoglobin in red blood cells that is glycosylated (attached to sugar) and is reported here as a percentage.
  percentage of glycosylated hemoglobin | 8.74 (1.41) | 8.81 (1.78) | 8.78 (1.60)

OUTCOME MEASURES:

1. Primary Outcome: Glucose Monitoring Adherence at Acute Outcome
Description: Medical adherence is a percent via the electronic monitoring using glucometer. This is a percent with a possible range of 0-100, with higher scores denoting better adherence.
Time Frame: Measured at Month 4
Measure: Mean (Standard Deviation); unit: percentage of glucose monitoring goal
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 42 | 45
percentage of glucose monitoring goal | 49.63 (4.66) | 79.79 (4.03)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; Multiple imputation was used to handle missing data; analyses are reported for the acute outcomes of glucose monitoring (i.e., 4 month); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; General linear model, controlling for baseline values; Mean Difference (Final Values) = 30.2, 95% CI 2-sided [17.37 to 42.9] — The Mean Difference was calculated as percent adherence to glucose monitoring for the CBT-AD Arm minus the adherence to glucose monitoring for the Enhanced Treatment as Usual Arm

2. Secondary Outcome: Glucose Control
Description: Hemoglobin A1C value at acute outcome. HbA1c is the number of hemoglobin in red blood cells that is glycosylated (attached to sugar) and is reported here as a percentage.
Time Frame: Month 4
Population: HbA1c as assessed by blood analysis
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 42 | 45
percentage of glycosylated hemoglobin | 8.58 (.16) | 7.86 (.16)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; Multiple imputation was used to handle missing data; results are reported for HbA1c at the acute outcome (i.e., 4 months); Test type: Superiority or Other; p = .001, ANCOVA; General linear model; Controlling for baseline values; Mean Difference (Final Values) = .72, 95% CI 2-sided [.29 to 1.15] — The Mean Difference was calculated as percent of HbA1c for the Enhanced Treatment as Usual Arm minus percent of HbA1c for the CBT-AD Arm

3. Primary Outcome: Percent Medication Adherence Via MEMS
Description: This is an electronic pill cap at the acute outcome assessment. This is a percent with a possible range of 0-100, higher scores indicating greater adherence
Time Frame: month 4
Population: Participants in each study arm
Measure: Mean (Standard Deviation); unit: Percentage of pills taken
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 42 | 45
Percentage of pills taken | 69.69 (3.72) | 90.37 (3.48)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; Analyses are reported for the acute outcomes of MEMs monitoring (4 month). Higher percentages represent better adherence; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 20.7, 95% CI 2-sided [10.22 to 31.14] — The Mean Difference was calculated as percent pill adherence via MEMs for the CBT-AD Arm minus the percent pill adherence for the Enhanced Treatment as Usual Arm

4. Primary Outcome: Clinician Rated Depression (MADRS) at the Acute Timepoint
Description: Depression as assessed by the Montgomery Asberg Depression Rating Scale (MADRS). This scale has a range of 0-60 with higher scores indicating greater depression severity.
Time Frame: month 4
Population: Participants in each arm
Measure: Mean (Standard Deviation); unit: units on a scale (MADRS)
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 42 | 45
units on a scale (MADRS) | 20.66 (1.52) | 14.22 (1.45)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; Analyses are reported for the acute outcomes of depression as assessed on the MADRS at acute outcome; Test type: Superiority or Other; p = .002, Mixed Models Analysis; General linear model, controlling for baseline values; Mean Difference (Final Values) = 6.22, 95% CI 2-sided [2.33 to 10.56] — The Mean Difference was calculated as MADRS unit scale for the CBT-AD Arm minus the MADRS unit scale for the Enhanced Treatment as Usual Arm

5. Primary Outcome: Depression on the CGI at Acute Outcome
Description: Clinical Global Impression is a scale from 1-7 with greater numbers meaning more severe depression
Time Frame: Month 4
Population: Participants in each study arm
Measure: Mean (Standard Deviation); unit: units on a scale - the CGI
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 42 | 45
units on a scale - the CGI | 3.17 (.20) | 2.44 (.21)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; Test type: Superiority or Other; p = .01, ANCOVA; using GLM; Mean Difference (Final Values) = .74, 95% CI 2-sided [.16 to 1.32] — The Mean Difference was calculated as CGI unit scale for the Enhanced Treatment as Usual Arm minus the CGI unit scale for the CBT-AD Arm

6. Other Pre Specified Outcome: Glucose Monitoring During Followup.
Description: This is a percent with a possible range of 0-100 with higher scores indicating better adherence. One Touch Ultra meters (LifeScan, Inc.) for daily glucose control provided frequency of self-monitoring, which when divided by the individualized goals from the nurse visits and multiplied by 100, yielded a percentage adherence score. This percentage adherence score was averaged at 4, 8, and 12 months between all participants in each arm, and those values were then averaged to give an overall percentage adherence score for each arm throughout the course of the study.
Time Frame: Aggregate of months 4,8,12
Measure: Mean (Standard Error); unit: percentage of glucose monitoring goal
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 42 | 45
percentage of glucose monitoring goal | 47 (5.5) | 69 (4.2)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; We hypothesized that differences in glucose monitoring adherence would continue to be superior in the CBT-AD condition compared to ETAU; Test type: Superiority or Other; p = .002, Mixed Models Analysis; Median Difference (Final Values) = 22.3, 95% CI 2-sided [8.6 to 36.1], Standard Error of Mean 7.0

7. Other Pre Specified Outcome: Percent Medication Adherence During Follow up
Description: Electronic pill cap adherence which indicates a percentage of doses taken. This percentage of doses taken was averaged at 4, 8, and 12 months between all participants in each arm, and those values were then averaged to give an overall percentage of doses taken for each arm throughout the course of the study.
Time Frame: Aggregate across 4,8,12 months
Measure: Mean (Standard Error); unit: percentage of doses taken
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 29 | 37
percentage of doses taken | 71 (4.5) | 87 (2.1)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; We hypothesized that the CBT-AD condition would maintain higher medication adherence over follow up compared to ETAU; Test type: Superiority or Other; p = .001, Mixed Models Analysis; Mean Difference (Final Values) = 16.3, 95% CI 2-sided [6.5 to 26.1], Standard Error of Mean 5.0

8. Other Pre Specified Outcome: Depression MADRS Over Follow up
Description: Independent (blind) assessor rating using the MADRS. This scale has a range of 0-60 with higher scores indicating greater depression severity. This depression score was averaged at 4, 8, and 12 months between all participants in each arm, and those values were then averaged to give an overall depression score for each arm throughout the course of the study.
Time Frame: Aggregate across 4,8,12 months
Measure: Mean (Standard Error); unit: Units on the MADRS scale
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 38 | 40
Units on the MADRS scale | 18.1 (1.5) | 15.1 (1.5)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; We hypothesized that the lower depression scores would remain in the CBT arm compared to ETAU over follow up; Test type: Superiority or Other; p = .16, Mixed Models Analysis; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-1.2 to 7.2], Standard Error of Mean 2.1

9. Other Pre Specified Outcome: Depression CGI
Description: Clinical Global Impression scale as rated by blinded interviewer. The CGI is a scale from 1-7 with greater numbers meaning more severe depression. This depression score was averaged at 4, 8, and 12 months between all participants in each arm, and those values were then averaged to give an overall depression score for each arm throughout the course of the study.
Time Frame: Aggregate 4,8,12 months
Measure: Mean (Standard Error); unit: Units on the CGI scle
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 38 | 42
Units on the CGI scle | 2.9 (.21) | 2.5 (.21)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; We hypothesized that depression scores would remain lower in the CBT-AD arm compared to the ETAU arm; Test type: Superiority or Other; p = .10, Mixed Models Analysis; Mean Difference (Final Values) = .48, 95% CI 2-sided [-.1 to 1.1], Standard Error of Mean .29

10. Other Pre Specified Outcome: Glucose Control Over Follow up
Description: Percent of HbA1c as assessed by blood analysis. HbA1c is the number of hemoglobin in red blood cells that is glycosylated (attached to sugar) and is reported here as a percentage. This percentage of HbA1c was averaged at 4, 8, and 12 months between all participants in each arm, and those values were then averaged to give an overall percentage of HbA1c for each arm throughout the course of the study.
Time Frame: Aggregate across 4,8,12 months
Population: HbA1c as assessed by blood analysis
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Number analyzed (Participants) | 38 | 40
percentage of glycosylated hemoglobin | 8.5 (2.2) | 7.9 (.19)
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual vs CBT-AD; We hypothesized that glucose control (HbA1C) would remain superior in the CBT-AD arm compared to the ETAU arm over follow up; Test type: Superiority or Other; p = .03, Mixed Models Analysis; Mean Difference (Final Values) = .63, 95% CI 2-sided [.6 to 1.2], Standard Error of Mean .29

ADVERSE EVENTS:
Arm/Group | Enhanced Treatment as Usual | CBT-AD
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/45
Other Adverse Events (participants affected / at risk) | 0/42 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No